CLINICAL TRIAL: NCT01698437
Title: MR-guided Ultrasound-Neurosurgery for the Treatment of Malignant Brain Tumors
Brief Title: Magnetic Resonance (MR) Guided Focused Ultrasound in the Treatment of Brain Tumors
Acronym: FUS-Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AG2010/026,ZH 2010-0543/3
Record Dates: First submitted 2012-05-29; First posted 2012-10-03 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Malignant Brain Tumors
Keywords: FUS; focused ultrasound; functional brain disorders; neuropathic pain; movement disorders; malignant of brain tumors
MeSH Terms: conditions — Neuralgia; Movement Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transcranial MR-Guided Focused Ultrasound for Brain Tumors (Other)
  Interventions: Device: Non-invasive intervention with focused ultrasound (ExAblate 4000)

INTERVENTIONS:
Device: Non-invasive intervention with focused ultrasound (ExAblate 4000) — Non-invasive brain intervention using MR-guided focused ultrasound
  Other Names: ExAblate 4000

SUMMARY:
Focused Ultrasound Focused ultrasound is an attractive method for non-invasive thermal ablation of soft tissue tumors. Treatment begins by acquiring a series of MR images of the target organ. The physician then identifies a target volume in the MR images and delineates the treatment contours on the images. Therapy planning software calculates the parameters required to effectively treat the defined target volume. During the treatment an ultrasound transducer generates and focuses ultrasound energy to a focal point, called a sonication. The sonication raises the tissue temperature within a well-defined region to a degree, which causes thermal coagulation. MR images acquired during sonication provide a quantitative, real-time temperature map of the target area to confirm the location of the sonication and the size of the coagulated region. The sonication process is repeated at multiple adjacent points to cover the entire prescribed treatment volume.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ages over 18 years old that give informed written consent to participate in study. Females in reproductive age have to provide a negative serum pregnancy test.
2. Patients with primary diagnosis (biopsy proven) of a malignant glioma or a recurrent glioma, that do not accept a conventional tumor resection or where a conventional tumor resection is not indicated according to both the neurosurgeon in charge and the neuro-oncology colloquium at the Kantonsspital Aarau.

   Or:

   Patients with a supratentorial brain metastasis of a malignant tumor, that do not accept a conventional tumor resection or where a conventional tumor resection is not indicated according to the neurosurgeon in charge and the neuro-oncology colloquium at the Kantonsspital Aarau.
3. The portion of the tumor to be treated during one intervention is less than 3.0 cm in diameter, corresponding to a volume of ca. 14 cc.

   If the total size of the tumor is larger than 3.0 cm in diameter then eventual complementing ablations will not be performed before 2 week after the first treatment.
4. The tumor to be treated is clearly defined and can be well distinguished from surrounding brain tissue.
5. The border of the targeted tumor volume has in all directions a distance of at least 2.5 cm from the inner table of the skull. Portions of the tumor that are not planned to be treated due to this safety margin will be marked.
6. Patients must have an ASA score 1-2, and a Karnofsky score 70-100

Exclusion Criteria:

All tumor Types

1. Clinical or neuroradiological signs of increased intracranial pressure.
2. Significantly increased vascularization of tumor in preoperative MR-angiogram or in digital subtraction angiography (DSA).
3. Tumor mass effect that causes midline shift or a shift of the third (3rd) ventricle of more than 5 mm, even after steroid therapy.
4. The border of the tumor portion to be treated is less then 5mm away from a main branch of a brain vessel, the venous sinuses, the pituitary gland or the cranial nerves.
5. The tumor is in immediate proximity to a cystic formation.
6. Recent (less than 2 weeks) intracranial hemorrhage.
7. Increased risk of bleeding: platelets < 100,000/mm3, INR > 1.3 or other coagulation disorders.
8. Tumors with presumably high risk of bleeding
9. Oral anticoagulant or thrombocyte aggregation suppression (e.g. ASS) that was not stopped at least 5 days before the intervention.
10. Contraindication for MR-exams, such as non-MR-compatible implants or cardiac pacemaker.
11. Clips and other implants in the sonication path or in the target area.
12. Operation implants such as dura patch, skull reconstruction with polymethylmethacrylate (PalacosTM), titan in the sonication path.
13. Infratentorial (i.e. cerebellar-) tumors.
14. Contraindications for MR-contrast agents or for steroid therapy
15. Allergy against local anesthesia.
16. Uncontrolled arterial hypertension.
17. Other life threatening diseases.
18. Severe uncontrolled systemic infection.
19. Hypersensitivity to contrast agents used in this study.
20. Severely impaired renal function (estimated glomerular filtration rate < 30 mL/min/1.73 m2) or under dialysis.
21. Inability to give informed written consent.
22. Alcohol or drug abuse.
23. Patients who are unreliable and will not appear for the follow up exams.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Lesion Size | 3 months
  Size of lesion in the tumor tissue for each sonication as a function of applied energy/temperature.
Patient Safety | 3 months
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Javier - Fandino, MD, Principal Investigator — Dept. of Neurosurgery, Kantonsspital Aarau, 5001 Aarau, Switzerland; Ernst - Martin, MD, Principal Investigator — Center for MR-Research, University Children's Hospital Zurich, Switzerland
Locations (1):
- MR-Center, University Children's Hospital, Zurich, Canton of Zurich, Switzerland